CLINICAL TRIAL: NCT07029529
Title: Phase 2 Dose-response Study of Apremilast in Women and Men With Alcohol Use Disorder
Brief Title: Dose-response Study of Apremilast in Women and Men With Alcohol Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2000040391; 2U54AA027989-06 (NIH)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Apremilast 60mg/day (Active Comparator): Apremilast 60mg/day. Administered orally twice daily at 8:00 AM and 8:00 PM while titrating to the full dose. Titration schedule: Day 1 10mg AM; Day 2 10mg AM, 10mg PM; Day 3 10mg AM, 20mg PM; Day 4 20mg AM, 20mg PM; Day 5 20 mg AM, 30mg PM; Day 6 30mg AM, 30mg PM. Once at steady state, administration is orally twice daily at 8:00 AM (30mg) and 8:00 PM (30mg).
  Interventions: Drug: Apremilast 60mg
- Apremilast 90mg/day (Active Comparator): Apremilast 90mg/day. Administered orally twice daily at 8:00 AM and 8:00 PM while titrating to the full dose. Titration schedule: Day 1 10mg AM; Day 2 10mg AM, 10mg PM; Day 3 10mg AM, 20mg PM; Day 4 20mg AM, 20mg PM; Day 5 20 mg AM, 30mg PM; Day 6 30mg AM, 30mg PM; Day 7 40mg AM, 30mg PM; Day 8 50mg AM, 30mg PM; Day 9 60mg AM, 30mg PM. Once at steady state, administration is orally twice daily at 8:00 AM (60mg) and 8:00 PM (30mg).
  Interventions: Drug: Apremilast 90mg
- Placebo (Placebo Comparator): Administered orally twice daily at 8:00 AM and 8:00 PM.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Apremilast 60mg — Apremilast 60mg/day
  Other Names: Otezla
  Arms: Apremilast 60mg/day
Drug: Apremilast 90mg — Apremilast 90mg/day
  Other Names: Otezla
  Arms: Apremilast 90mg/day
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
For this protocol, the investigators plan to collect data to evaluate apremilast (60mg/day or 90mg/day) vs placebo in adults with Alcohol Use Disorders (AUD).

DETAILED DESCRIPTION:
This human laboratory study is a Phase 2 double-blind, placebo-controlled, dose-response, parallel group design which will compare apremilast (90mg/day vs 60mg/day) to placebo in non-treatment seeking adults meeting criteria for DSM 5 alcohol use disorders (n=120, 40 per cell, 50% females).

Eligibility screening consists of an intake session and a physical exam. Subjects meeting eligibility criteria will be assigned to apremilast (90mg/day or 60mg/day) or placebo. Titration to steady state medication levels occur over 9 days (Day 1-9). Subjects will then complete three laboratory sessions (Days 10-24). During each laboratory session, personalized imagery (within-subject factor, either stress or stimulation or neutral, order counterbalanced) will precede a 2-hour alcohol self-administration period. Participants will remain on study medication for a 30-day period, during which naturalistic drinking will be evaluated.

No taper medication is needed. Following the discontinuation of medication (Day 30), participants will be assessed for an additional 1-month period.

Adverse events are evaluated at each study appointment and will be tabulated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65.
2. Able to read and write English.
3. Meets DSM-5 criteria for current (past 6 months) AUD.
4. Drinking criteria: males - drinks > 14 drinks per week and exceeds 4 drinks per day at least twice per week; females - drinks > 7 drinks per week and exceeds 3 drinks per day at least twice per week. They must meet drinking criteria during a consecutive 30-day period prior to baseline.
5. Laboratory sessions will be scheduled such that subjects will not have major responsibilities on the following day which might limit drinking during the self-administration session (e.g., job interview, exam).
6. Able to take oral medications and willing to adhere to medication regimen.
7. Provision of signed and dated informed consent form
8. Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

1. Subjects with any significant current medical conditions (neurological, cardiovascular, endocrine, thyroid, renal, liver), seizures, delirium or hallucinations, or other unstable medical conditions, including HIV.
2. Current DSM-5 substance use disorder (other than AUD or tobacco use disorder).
3. A positive test result at intake appointment on urine drug screens conducted for illicit drugs.
4. Past 30-day use of psychoactive drugs may be included at the discretion of the study MD as long as the concurrent treatment does not compromise the study integrity by virtue of its type, duration, or intensity.
5. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or her partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD).
6. Suicidal, homicidal, or evidence of current (past 6 months) mental illness such as schizophrenia, bipolar disorder or major depression, or anxiety disorders.
7. Only one member per household can participate in the study.
8. Specific exclusions for administration of apremilast not already specified include: known hypersensitivity to apremilast; cytochrome P450 enzyme inducers (e.g., rifampin, phenobarbital, carbamazepine, phenytoin).
9. Drugs that may influence study outcomes (e.g., disulfiram, naltrexone, acamprosate, anticonvulsants).
10. Subjects likely to exhibit clinically significant alcohol withdrawal during the study. We will exclude subjects who a) have a history of perceptual distortions, seizures, delirium, or hallucinations upon withdrawal, or b) have a score of > 8 on the Clinical Institute Withdrawal Assessment scale at intake appointments.
11. Subjects who have taken any investigational drug within 4 weeks immediately preceding admission to the study period.
12. Participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current application.
13. Individuals who are currently in treatment for drinking or who have attempted to quit drinking within the past 3 months in order to exclude participants seeking treatment.
14. Individuals with a history of serious withdrawal, and individuals who have repeatedly undergone alcohol detoxification.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | Lab Sessions (Days 10, 17 & 24)
  For the ad-libitum drinking sessions (120 mins), the primary outcome variable will be calculated as percent milliliters consumed = number of milliliters consumed/total amount available.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No